CLINICAL TRIAL: NCT04786639
Title: Comparison of Surgical Fixation and Non-Operative Management Outcomes in Proximal Humerus Fractures
Brief Title: Surgical Fixation and Non-Operative Management Outcomes in Proximal Humerus Fractures
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assistant Prof., Istanbul University - Cerrahpasa
Other Study IDs: IUC1
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Fixation Group: Open reduction with deltopectoral incision and humeral osteosynthesis with anatomic plates and screws will be performed for surgical fixation.
- Non-Operative Group: Non-surgical treatment will be performed with sling immobilization.

SUMMARY:
The management of proximal humerus fractures (PHFs) remains a significant challenge in orthopaedics. The acute treatment options for PHFs are numerous and are typically guided by the fracture pattern and functional demands of the patients. The most commonly used methods include non-operative management with a sling or surgical fixation. Although non-surgical treatment is a reasonable treatment option for the majority of humerus fractures, there is an increasing interest in surgical intervention. There are no evidence-based treatment recommendations, thus permitting large local variation in treatment preferences.

There are a number of studies in the literature about how outcome measures of the patients after PHFs management change, but these results generally compare functional results before and after treatment. Misra et al. stated that conservatively managed patients with PHFs have more pain and a poorer range of motion than those managed by either fixation or arthroplasty, while cochrane review stated that surgery is not superior to nonsurgical treatment in most proximal humerus fractures. Jayakumar et al. determined that kinesiophobia is one of the strongest predictors of functional limitation and recovery from a PHF is enhanced by overcoming fears of movement or reinjury within a week after injury.

There is no clear knowledge regarding how the surgical or conservative management used in the management of PHF affects the early results of assessment parameters. The aim of this study was to compare early results of surgical fixation versus non-operative management outcomes in patients with proximal humerus fractures.

DETAILED DESCRIPTION:
Voluntary patients who have been diagnosed with proximal humerus fracture and managed by surgical or conservative will be included in the study.

Patients with stabilization after proximal humerus fracture with surgical fixation will be considered as the Surgery group, and patients treated with non-surgical treatment with sling immobilization will be considered as the Conservative group. Signed voluntary consent will be obtained from participants. Patients having surgical fixation or nonoperative management will be assessed for kinesiophobia, pain, range of motion, functional status, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Stabilization after proximal humerus fracture with surgical fixation (post-op 3-6 weeks) or non-surgical treatment with sling immobilization (callus formation on radiography).
* Volunteer

Exclusion Criteria:

* Malunion tubercle majus,
* Advanced osteoporosis,
* Avascular necrosis of the humeral head,
* Presence of neurological and rheumatologic disease,
* Recurrent infection and open wound-incision in the region,
* Communication problems

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with proximal humerus fracture who come to the orthopedic clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia | Baseline
  Tampa kinesiophobia scale will be used for determining of kinesiophobia or fear of movement.The Tampa Scale for Kinesiophobia is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. The score varies between 17 and high scores indicate an increasing degree of kinesiophobia.

SECONDARY OUTCOMES:
Shoulder Pain | Baseline
  A Visual Analogue Scale will be used for pain of rest, night and activity. It is a scale measuring the distance (mm) on the 10-cm line between the "no pain" (0) and and " worst pain (10).
Range of Motion | Baseline
  Shoulder flexion, extension, external and internal rotation will be measured by using digital goniometer. It is a reliable and valid tool for measuring shoulder range of motion in individuals with healthy shoulders. Increasing the degree is considered as an improvement in the range of motion.
Functional Status | Baseline
  The Disabilities of the Arm, Shoulder and Hand questionnaire will be used for measuring of self-rated upper-extremity disability and symptoms. The scale score ranging is from 0 (no disability) to 100 (most severe disability).
Quality of Life of the patients | Baseline
  The quality of life will be assessed by using 36-Item Short Form Survey. The survey has eight sub scaled scores; vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. Scores range from 0 - 100 and higher scores shows less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Ayşe Alpözgen, Küçükçekmece, Istanbul, Turkey (Türkiye)